Evaluation of an Expectancy Challenge Intervention for Food and Alcohol Disturbance (FAD) Among College Students

NCT06810414

Document Date: 12/19/2024

# Consent for Participating in Research Eating, Alcohol, and Other Health-Related Behaviors Among College Students

## **Study Contact**

Katherine Berry, M.S., Principal Investigator Clinical Psychology Doctoral Student Department of Psychology, University of Wyoming Email: kberry11@uwyo.edu

Alison Looby, Ph.D., Faculty Supervisor Professor Department of Psychology, University of Wyoming Email: alooby@uwyo.edu

# **Purpose of this Research**

The purpose of this research is to learn more about eating, alcohol, and other health-related behaviors on college campuses. You are being invited to participate in this study because you are a college student between the ages of 18 and 25.

## **Description of the Research Study**

This study requires one in-person group-based laboratory visit, which should take approximately two hours to complete, and one online follow-up survey which should take about 15-20 minutes to complete. During the in-person laboratory visit, you will complete questionnaires, participate in discussions with other group members, and engage in written exercises about eating, alcohol use, and other health-related behaviors. The researcher will explain the questionnaires and discussions and writing exercises before you complete them, and you will have the opportunity to ask questions. During the online follow-up survey, you will complete questionnaires remotely from a device of your choosing. You will complete these questionnaires one-month following your initial in-person lab visit.

## Risks

There are some minor risks involved in participating in this study. During completion of questionnaires and the discussions and writing exercises, you may become uncomfortable, anxious, or experience feelings of shame when learning about, discussing, or writing about eating, alcohol use, and other health-related behaviors. Since you may be providing our laboratory with sensitive information about your alcohol use, there is a very minimal chance that this information could be exposed to outside parties, including law enforcement. We are taking steps to ensure that this does not happen. Your name will never be associated with the data you provide our laboratory. Upon all completion of data collection related to this study, all identifiable information will be deleted. In addition, given the group-based nature of this study, there is a potential risk that participants might share information disclosed by others during group activities. However, we hope to minimize this risk by establishing clear group rules at the outset and asking participants to verbally agree not to disclose any information discussed during the study, including information discussed by the other participants or tell others about the other individuals who participated.

#### **Benefits:**

Participation in this study may increase your awareness of your eating, alcohol use, and other health-related behaviors. It is also possible that you will not receive any benefits from this research. Although you may not receive direct benefit from your participation, others may ultimately benefit from the knowledge obtained from this research regarding better understanding of health-related behaviors on college campuses.

#### **Compensation:**

For those participating via Sona, you will receive 2 Sona credits to be applied to a psychology course at the University of Wyoming for participating in the first study visit. For those recruited from outside of Sona, you will receive a \$40 gift card for participating in the first study visit. Should you withdraw from the study prior to its completion, you will receive compensation commensurate with the amount of time you participated prior to withdrawal. All participants will receive a \$20 gift card for completing the one-month follow-up survey. If you do not complete the survey within 30 days of receiving the initial email with the survey link, you will not be compensated. Further, if you start completing the follow-up survey, but do not finish it, you will not be compensated.

#### **Confidentiality**

All information obtained in this study will be treated confidentially and privately to the extent permitted by law. Data from your pre-screening survey as well as documentation of your participation in the study and your email address and name, which will be used for follow-up purposes, will be stored on the password-protected computer in our laboratory. All records from the study are stored in locked file cabinets and on password protected computers. All data that you provide in the study visits will be identified by subject numbers rather than name. Only the researchers will have access to these records. The information obtained in this study will be used for research investigational purposes and your name will never be publicly disclosed at any time. You will not be identifiable in any publication that may arise from this research. Any information that is obtained in this study and that can be identified with you will remain confidential and will be disclosed only with your permission or as required by law. Records will be kept in our laboratory for a minimum of 3 years and then destroyed.

## **Compensation for Injury**

If you should suffer any injury as a result of participation, please understand that no provision has been made to provide treatment for injury or any other financial compensation. In the unlikely event that you become ill or injured as a direct result of participating in this study, the University of Wyoming has no funds budgeted for compensation for injury, damages, or other expenses. However, you should report any such injury or adverse emotional reactions to the principal investigator, Katherine Berry, M.S. (email: <a href="mailto:kberry11@uwyo.edu">kberry11@uwyo.edu</a>, phone: 307-314-2669) or the faculty supervisor, Dr. Looby (email: <a href="mailto:alooby@uwyo.edu">alooby@uwyo.edu</a>, phone: 307-314-2314).

# **Voluntary Participation:**

Your participation in this project is voluntary. Even after you agree to participate in the research, you may decide to discontinue the study at any time without penalty or loss of benefits to which you may otherwise have been entitled, simply by informing the researcher that you no longer wish to participate. You may choose not to answer any questions and may refuse to complete any portions of the research you do not wish to for any reason. Your refusal to participate will not have any effect on your present or future relationship with the University of Wyoming.

## **Additional Information:**

Direct questions or concerns regarding this study can be directed to the principal investigator, Katherine Berry, M.S. (email: <a href="kberry11@uwyo.edu">kberry11@uwyo.edu</a> phone: 307-314-2669) or the faculty supervisor of the research study, Alison Looby, PhD (email: <a href="alooby@uwyo.edu">alooby@uwyo.edu</a> phone: 307-314-2314). If you have any questions regarding your rights as a research subject, or if you have any concerns or complaints about the research, you may contact the University of Wyoming Institutional Review Board at (307) 766-5320.

# Before you agree to the provisions of this document:

I have read the consent form and made sure that I have a thorough understanding of the research study. I understand that I am not waiving any legal rights by signing this form. If I decide to participate in this research study, I can be provided with a copy of this document for my own personal records.

| Name (please print): | Date: | |
|---|---|---|
| Signature: | | |
| Do you agree to be contacted via text | message regarding follow-up participation in this | study |
| Yes (please provide your cell pho | ne number): | |
| No | | |